



## PREFECTUS STUDY: Informed Consent Form

Please initial each box.

| 1. | I confirm that I have read a | nd understood the inform | ation sheet dated | | | |
|---|---|---|---|---|---|---|
| | (Version) for the above study and that I have had the | | | | | |
| | opportunity to ask question | ns. | | | | |
| 2. | I understand that my participation in the study is voluntary and that I am | | | | | |
| | free to withdraw at any time without giving any reason. This will not | | | | | |
| | affect my treatment in any way. | | | | | |
| 3. | . I agree to take part in the above study. | | | | | |
| 4. | I give permission for my GP to be informed about my participation in the study. | | | | | |
| 5. | I give permission for my hospital clinical record to be reviewed by the research team for this project. | | | | | |
| 6. | I give permission for transferring of all of my research study data in anonymised form onto a database to be stored within Cardiff School of Sport, Cardiff Metropolitan University | | | | | |
| 7. | I give permission to contact me by telephone 6-12 months after the final study visit to ask some questions about my health and general condition. | | | Yes | No | |
| | | | | | | - |
| Name of participant | | Date | Signati | Signature | | |
| Name of person taking consent | | Date | Signati | Signature | | - |
| (if different from researcher) | | | | | | |
| | | Date | Signati | Signature | | |